CLINICAL TRIAL: NCT03806075
Title: Molecular Typing and Precise Prevention and Treatment of Peutz-Jeghers Syndrome
Brief Title: Study of Accurate Diagnosis and Treatment of Peutz-Jeghers Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yiqi Du (Other)
Responsible Party: Sponsor-Investigator, Yiqi Du, Professor, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017JZ13
Record Dates: First submitted 2019-01-13; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Peutz-Jeghers Syndrome
Keywords: Second generation gene sequencing, gut microbiota, Gastrointestinal polyp syndrome
MeSH Terms: conditions — Peutz-Jeghers Syndrome

STUDY DESIGN:
Intervention Model Description: All patients with Peutz-Jeghers were enrolled and accepted second generation gene sequencing. Then all patients allocated into gene mutation group and no gene mutation group according to if the cases accompany with gene mutation of STK11.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peutz-Jeghers patients (Experimental): All Peutz-Jeghers patients meet the clinical criteria
  Interventions: Behavioral: Second generation sequencing; Behavioral: 16s rRNA gene sequencing
- Health persons (Placebo Comparator): Those without Peutz-Jeghers syndrome
  Interventions: Behavioral: 16s rRNA gene sequencing

INTERVENTIONS:
Behavioral: Second generation sequencing — Firstly, all Peutz-Jeghers patients accept second generation gene sequencing with their blood specimen
  Arms: Peutz-Jeghers patients
Behavioral: 16s rRNA gene sequencing — Secondly, All patients and Health persons accepted 16s rRNA gene sequencing with their feces specimen

SUMMARY:
The mutation of STK11 has been regcognized to be the major cause of Peutz-Jeghers syndrome (PJS).The aim of this study was to confirm the mutation rate of gene associated with gastrointestinal malignancies,including STK11, APC,PMS1,et al. Furtherly, the investigators analyze the association of STK11 with gut microbiota.

DETAILED DESCRIPTION:
All patients diagnosed as PJS were enrolled and accepted second generation gene sequencing with their blood specimens. Then all patients allocated into gene mutation group and no gene mutation group according to if the cases accompany with gene mutation of STK11.Also, health persons were enrolled and a case controlled study will be carried out.All patients and health persons accepted 16s rRNA sequencing with their feces specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with ages from 18-70 years old.
2. Subject diagnosed with Peutz-Jeughers syndrome.
3. Subject without hypertension, diabetes and other gastrointestinal diseases.
4. The consent form has been signed.

Exclusion Criteria:

1. Subject is younger than 18 years or older than 70 years.
2. Subject with hypertension,diabetes and other gastrointestinal diseases.
3. Subject taken or adminstered medicine associated with digestive function during latest 1 month.
4. Pregnant women.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Mutation of gene associated with Peutz-Jeghers syndrome | 2 years
  Mutation of gene associated with Peutz-Jeghers syndrome, including STK11, APC,PMS1,PMS2 et al.

SECONDARY OUTCOMES:
Intestinal microbiota of patients with PJS | 1year
  Identify the variation of intestinal microbiota of patients with PJS

OTHER OUTCOMES:
The association of STK11 with intestinal microbiota of patients with PJS | 1 year
  The association of STK11 with intestinal microbiota of patients with PJS

CONTACTS AND LOCATIONS:
Overall Officials: Yiqi Du, Ph.D., Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No